CLINICAL TRIAL: NCT02598752
Title: Feasibility and Safety of Functional Performance Testing in Patients Undergoing Hematopoietic Cell Transplantation
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 15-274
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Hematological Malignancy; Leukemia; Lymphoma; Myeloma
Keywords: functional performance testing; exercise fitness testing; 15-274
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Hematologic Neoplasms; Leukemia; Lymphoma; Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- functional performance testing: This observational study will evaluate the feasibility and safety of functional performance testing in patients undergoing HCT. In addition to standard of care procedures, participants will undergo a CPET with a rest and stress echo, pulmonary function, and patient reported outcome questionnaires within 30 days of HCT.
  Interventions: Other: Symptom-limited cardiopulmonary exercise test (CPET); Other: Resting assessment of cardiac function by echocardiography; Other: Post-exercise assessment of cardiac function by echocardiography; Other: Pulmonary function; Behavioral: Patient-reported outcomes questionnaire

INTERVENTIONS:
Other: Symptom-limited cardiopulmonary exercise test (CPET)
Other: Resting assessment of cardiac function by echocardiography
Other: Post-exercise assessment of cardiac function by echocardiography
Other: Pulmonary function
Behavioral: Patient-reported outcomes questionnaire

SUMMARY:
The purpose of this study is to see if exercise fitness testing is feasible and safe in persons over 21 years of age who have been diagnosed with a hematological malignancy and are scheduled to undergo a hematopoietic stem cell transplant (HCT). Assessments in this study will look at the capacity of the body before transplantation to see if these measures can help predict how patients do after transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MSK histologically confirmed hematologic malignancy
* Scheduled for autologous or allogenic HCT at MSKCC
* ≥21 years old
* ECOG performance status of 0 or 1
* Completion of baseline CPET
* Willing to comply with protocol related procedures

Exclusion Criteria:

* Any of the following absolute contraindications to cardiopulmonary exercise testing

  * Acute myocardial Infarction (within 3-5 days of any planned study procedures)
  * Unstable angina
  * Uncontrolled arrhythmia causing symptoms or hemodynamic compromise
  * Recurrent syncope
  * Active endocarditis
  * Acute myocarditis or pericarditis
  * Symptomatic severe aortic stenosis
  * Uncontrolled heart failure
  * Acute pulmonary embolus or pulmonary infarction within 3 months of any planned study procedures
  * Thrombosis of lower extremities
  * Suspected dissecting aneurysm
  * Uncontrolled asthma
  * Pulmonary edema
  * Respiratory failure
  * Acute non-cardiopulmonary disorders that may affect exercise performance or be aggravated by exercise (i.e., infection, renal failure, thyrotoxicosis)
  * Presence of any other concurrent, actively treated malignancy;
  * History of any other malignancy treated within the past 3 years (other than non-melanoma skin cancer);
  * Room air desaturation at rest ≤85%
  * Mental impairment leading to inability to cooperate

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potentially eligible will be identified through and recruited from the Adult Bone Marrow Transplantation clinics at MSK.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
VO2peak | 1 year
  is a measure determined by the CPET

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Scott, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/